CLINICAL TRIAL: NCT00300131
Title: Bioabsorbable Vascular Solutions First in Man Clinical Investigation: A Clinical Evaluation of the Bioabsorbable Vascular Solutions Everolimus Eluting Coronary Stent System (BVS EECSS) in the Treatment of Patients With Single de Novo Native Coronary Artery Lesions
Brief Title: ABSORB Clinical Investigation, Cohort A (ABSORB A) Everolimus Eluting Coronary Stent System Clinical Investigation
Acronym: ABSORB A
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 05-370
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Bioabsorbable; Coronary Stent; Everolimus; drug eluting stents; stents; angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Bioabsorbable Vascular Solutions (BVS) Everolimus Eluting Coronary Stent System
  Interventions: Device: Bioabsorbable Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: Bioabsorbable Everolimus Eluting Coronary Stent — Bioabsorbable drug eluting stent implantation stent in the treatment of coronary artery disease
  Other Names: BVS

SUMMARY:
Prospective, open-labeled First in Man Clinical Investigation enrolling patients with visually estimated nominal vessel diameter of 3.0 mm receiving a single 3.0 x 12 mm or 3.0 x 18 mm BVS EECSS containing 98 microgramme per cm² of surface area.

DETAILED DESCRIPTION:
* Prospective, open-labeled Clinical Investigation enrolling patients with visually estimated nominal vessel diameter of 3.0 mm and lesion length ≥ 8 mm receiving a single 3.0 x 12 mm BVS Everolimus Eluting CSS containing 98 microgramme per cm² of surface area. Lesion length will be expanded to≥ 14 mm in length by visual estimation when 3.0 x 18 mm stent is available.
* Angiographic, Intravascular Ultrasound (IVUS), Intravascular Ultrasound- virtual histology (IVUS-VH) and Palpography follow-up will be carried out in all patients at 180 days and 2 years following the index procedure
* Optical Coherence Tomography (OCT) follow-up at 180 days and 2 years will be carried out in a subset of up to 10 patients in Cohorts A and B respectively who are enrolled in pre-determined clinical site(s)
* Multi-slice Spiral Computed Tomography (MSCT) is an optional procedure which may be carried out at 18 months post procedure and again between 4 and 5 year follow up.
* Additionally, coronary vasomotion test may be done at 2 years post procedure

Single patient Cohort of 30.

Pipeline products. Currently in development at Abbott Vascular. Not available for sale.

ELIGIBILITY:
Inclusion Criteria:

Target lesion must be located in a native epicardial vessel with visually estimated nominal vessel diameter of 3.0 mm

* Target lesion must measure less/equal 8 mm in length by visual estimation for 3.0 x 12 mm, expanded to less/equal 14 mm in length by visual estimation when 3.0 x 18 mm stent is available
* The target lesion(s) must be in a major artery or branch with a visually estimated stenosis of > 50% and < 100% with a TIMI flow of greater/equal 1
* Non-Clinical Investigation, percutaneous intervention for lesions in a non-target vessel is allowed if done more/equal 90 days prior to or if planned to be done 6 months after the index procedure
* Non-Clinical Investigation, percutaneous intervention for lesions in the target vessel is allowed if done > 6 months prior to or if planned to be done 6 months after the index procedure

Exclusion Criteria:

* Located within an arterial or saphenous vein graft or distal to a diseased (defined as vessel irregularity per angiogram and > 20% stenosed lesion by visual estimation) arterial or saphenous vein graft
* Lesion involving a bifurcation greater/equal 2 mm in diameter and ostial lesion > 40% stenosed by visual estimation or side branch requiring predilatation
* Total occlusion (TIMI flow 0), prior to wire passing
* The target vessel contains visible thrombus
* Another clinically significant lesion is located in the same epicardial vessel (including side branch) as the target lesion
* Patient has received brachytherapy in any epicardial vessel (including side branches)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Ischemia Driven MACE | at 30, 180, 270 days, and 1, 2, 3, 4, 5 years;
Ischemia driven Target Vessel Failure (TVF) | at 30, 180, 270 days, and 1, 2, 3, 4, 5 years;
Acute success (clinical device and clinical procedure) | Acute
Ischemia Driven Target Lesion Revascularization (TLR) | at 30, 180, 270 days and 1, 2, 3, 4, 5 years;
Ischemia Driven Target Vessel Revascularization (TVR) | at 30, 180, 270 days and 1, 2, 3, 4, 5 years

SECONDARY OUTCOMES:
In-stent Late Loss(LL) | at 180 days and 2 years
In-segment LL | at 180 days and 2 years
Proximal LL (proximal defined as within 5 mm of tissue proximal to stent placement) | at 180 days and 2 years
Distal LL (distal defined as within 5 mm of tissue distal to stent placement) | at 180 days and 2 years
In-stent and in-segment Angiographic Binary Restenosis (ABR) rate | at 180 days and 2 years
In-stent % Volume Obstruction (VO) | at 180 days and 2 years
Persisting incomplete apposition, late incomplete apposition, aneurysm, thrombus, persisting dissection | at 180 days and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Ormiston, MD, Principal Investigator — Auckland City Hospital; Patrick Serruys, MD, Principal Investigator — Erasmus University Thorax Center
Locations (4):
- Skejby Sygehus, Aarhus, Denmark
- Erasmus University Thorax Center, Rotterdam, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- University Hospital, Krakow, Poland

REFERENCES:
- [Background] Ormiston JA, Webster MW, Armstrong G. First-in-human implantation of a fully bioabsorbable drug-eluting stent: the BVS poly-L-lactic acid everolimus-eluting coronary stent. Catheter Cardiovasc Interv. 2007 Jan;69(1):128-31. doi: 10.1002/ccd.20895. PMID 17139655
- [Background] TCT Daily: ABSORB: bioabsorbable coronary stents successfully and safely deployed. J Interv Cardiol. 2007 Feb;20(1):36-7. doi: 10.1111/j.1540-8183.2007.00235.x. No abstract available. PMID 17300400
- [Result] Tanimoto S, Serruys PW, Thuesen L, Dudek D, de Bruyne B, Chevalier B, Ormiston JA. Comparison of in vivo acute stent recoil between the bioabsorbable everolimus-eluting coronary stent and the everolimus-eluting cobalt chromium coronary stent: insights from the ABSORB and SPIRIT trials. Catheter Cardiovasc Interv. 2007 Oct 1;70(4):515-23. doi: 10.1002/ccd.21136. PMID 17503509
- [Result] Ormiston JA, Serruys PW, Regar E, Dudek D, Thuesen L, Webster MW, Onuma Y, Garcia-Garcia HM, McGreevy R, Veldhof S. A bioabsorbable everolimus-eluting coronary stent system for patients with single de-novo coronary artery lesions (ABSORB): a prospective open-label trial. Lancet. 2008 Mar 15;371(9616):899-907. doi: 10.1016/S0140-6736(08)60415-8. PMID 18342684
- [Result] Serruys PW, Ormiston JA, Onuma Y, Regar E, Gonzalo N, Garcia-Garcia HM, Nieman K, Bruining N, Dorange C, Miquel-Hebert K, Veldhof S, Webster M, Thuesen L, Dudek D. A bioabsorbable everolimus-eluting coronary stent system (ABSORB): 2-year outcomes and results from multiple imaging methods. Lancet. 2009 Mar 14;373(9667):897-910. doi: 10.1016/S0140-6736(09)60325-1. PMID 19286089
- [Result] Garcia-Garcia HM, Gonzalo N, Pawar R, Kukreja N, Dudek D, Thuesen L, Ormiston JA, Regar E, Serruys PW. Assessment of the absorption process following bioabsorbable everolimus-eluting stent implantation: temporal changes in strain values and tissue composition using intravascular ultrasound radiofrequency data analysis. A substudy of the ABSORB clinical trial. EuroIntervention. 2009 Jan;4(4):443-8. doi: 10.4244/eijv4i4a77. PMID 19284065
- [Result] Tanimoto S, Bruining N, van Domburg RT, Rotger D, Radeva P, Ligthart JM, Serruys PW. Late stent recoil of the bioabsorbable everolimus-eluting coronary stent and its relationship with plaque morphology. J Am Coll Cardiol. 2008 Nov 11;52(20):1616-20. doi: 10.1016/j.jacc.2008.08.024. PMID 18992650
- [Result] Bruining N, Tanimoto S, Otsuka M, Weustink A, Ligthart J, de Winter S, van Mieghem C, Nieman K, de Feyter PJ, van Domburg RT, Serruys PW. Quantitative multi-modality imaging analysis of a bioabsorbable poly-L-lactic acid stent design in the acute phase: a comparison between 2- and 3D-QCA, QCU and QMSCT-CA. EuroIntervention. 2008 Aug;4(2):285-91. doi: 10.4244/eijv4i2a49. PMID 19110796
- [Result] Ormiston JA, Serruys PW. Bioabsorbable coronary stents. Circ Cardiovasc Interv. 2009 Jun;2(3):255-60. doi: 10.1161/CIRCINTERVENTIONS.109.859173. No abstract available. PMID 20031723
- [Result] Macaya C, Moreno R. Bioabsorbable drug-eluting stents: the future of coronary angioplasty? Nat Clin Pract Cardiovasc Med. 2008 Oct;5(10):598-9. doi: 10.1038/ncpcardio1306. Epub 2008 Aug 5. PMID 18679382
- [Result] Onuma Y, Piazza N, Ormiston JA, Serruys PW. Everolimus-eluting bioabsorbable stent--Abbot Vascular programme. EuroIntervention. 2009 Dec 15;5 Suppl F:F98-F102. doi: 10.4244/EIJV5IFA17. No abstract available. PMID 22100687
- [Result] Oberhauser JP, Hossainy S, Rapoza RJ. Design principles and performance of bioresorbable polymeric vascular scaffolds. EuroIntervention. 2009 Dec 15;5 Suppl F:F15-22. doi: 10.4244/EIJV5IFA3. PMID 22100671
- [Result] Onuma Y, Serruys PW, Perkins LE, Okamura T, Gonzalo N, Garcia-Garcia HM, Regar E, Kamberi M, Powers JC, Rapoza R, van Beusekom H, van der Giessen W, Virmani R. Intracoronary optical coherence tomography and histology at 1 month and 2, 3, and 4 years after implantation of everolimus-eluting bioresorbable vascular scaffolds in a porcine coronary artery model: an attempt to decipher the human optical coherence tomography images in the ABSORB trial. Circulation. 2010 Nov 30;122(22):2288-300. doi: 10.1161/CIRCULATIONAHA.109.921528. Epub 2010 Oct 25. PMID 20975003
- [Derived] Onuma Y, Dudek D, Thuesen L, Webster M, Nieman K, Garcia-Garcia HM, Ormiston JA, Serruys PW. Five-year clinical and functional multislice computed tomography angiographic results after coronary implantation of the fully resorbable polymeric everolimus-eluting scaffold in patients with de novo coronary artery disease: the ABSORB cohort A trial. JACC Cardiovasc Interv. 2013 Oct;6(10):999-1009. doi: 10.1016/j.jcin.2013.05.017. PMID 24156961
- [Derived] Brugaletta S, Gogas BD, Garcia-Garcia HM, Farooq V, Girasis C, Heo JH, van Geuns RJ, de Bruyne B, Dudek D, Koolen J, Smits P, Veldhof S, Rapoza R, Onuma Y, Ormiston J, Serruys PW. Vascular compliance changes of the coronary vessel wall after bioresorbable vascular scaffold implantation in the treated and adjacent segments. Circ J. 2012;76(7):1616-23. doi: 10.1253/circj.cj-11-1416. Epub 2012 Apr 24. PMID 22531596
- [Derived] Dudek D, Onuma Y, Ormiston JA, Thuesen L, Miquel-Hebert K, Serruys PW. Four-year clinical follow-up of the ABSORB everolimus-eluting bioresorbable vascular scaffold in patients with de novo coronary artery disease: the ABSORB trial. EuroIntervention. 2012 Jan;7(9):1060-1. doi: 10.4244/EIJV7I9A168. PMID 21959320